CLINICAL TRIAL: NCT01370278
Title: Clearance Of Mucus In Stents (COMIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2010-0990; NCI-2011-01119 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Lung Neoplasms; Respiratory Failure; Pneumonia; Acute Coronary Syndromes; Unstable Angina; Myocardial Infarction; Cardiac Arrhythmia; Thromboembolic Disease
Keywords: Central airway obstruction; lumen obstruction; Sodium bicarbonate; Baking soda; Normal saline; Salt water; Airway stents; Bronchoscopy; mucus obstruction
MeSH Terms: conditions — Lung Neoplasms; Respiratory Insufficiency; Pneumonia; Acute Coronary Syndrome; Angina, Unstable; Myocardial Infarction; Arrhythmias, Cardiac; Thromboembolism | interventions — Saline Solution; Fluoridation; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): Normal saline sprayed into stent/airway tubes then suctioned out through bronchoscope.
  Interventions: Other: Normal Saline
- Sodium Bicarbonate (Active Comparator): Sodium bicarbonate sprayed into stent/airway tubes then suctioned out through bronchoscope.
  Interventions: Other: Sodium Bicarbonate

INTERVENTIONS:
Other: Normal Saline — Normal saline administered in stent/airway tubes under direct visualization via the bronchoscope.
  Other Names: Salt water
  Arms: Normal Saline
Other: Sodium Bicarbonate — 4.2% bicarbonate solution mixed with equal volume of sterile water administered into stent/airway tubes under direct visualization via the bronchoscope.
  Other Names: Baking soda
  Arms: Sodium Bicarbonate

SUMMARY:
The goal of this clinical research study is to compare the effects of sodium bicarbonate to normal saline when used for clearing mucus blockage in patients with airway stents.

DETAILED DESCRIPTION:
Study Agents:

Sodium bicarbonate is also called baking soda. In this study it will be mixed with water.

Normal saline is a salt water solution.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. The study doctor will use either sodium bicarbonate or normal saline during your bronchoscopy to clear mucus from your stent:

* If you are in Group 1, the study doctor will use sodium bicarbonate. The amount of sodium bicarbonate in the solution will be the same for all patients in Group 1.
* If you are in Group 2, the study doctor will use normal saline.

You will have an equal chance of being assigned to either group. Neither you nor the study staff can choose the group you will be in, and neither you nor your doctor will know if you are receiving sodium bicarbonate or normal saline. However, if needed for your safety, the study staff will be able to find out what you are receiving.

If you have more than 1 stent, only 1 of your stents will be checked for clearance of mucus in this study. However, all stents will be cleared of mucus if needed.

As part of your standard of care, you will have photographs and videos taken before and after your bronchoscopy. You will sign a separate consent form for your bronchoscopy. Your complete medical history will also be recorded.

For the bronchoscopy, you will be given drugs to help you relax, and then a local anesthetic will be sprayed into your nose and throat to numb those areas. A slim, flexible tube with a light will be placed through your nose or mouth and into your airway tubes.

If you are in Group 1, a small amount of sodium bicarbonate will be sprayed into your stent/airway tubes and then suctioned out through the bronchoscope.

If you are in Group 2, a small amount of normal saline will be sprayed into your stent/airway tubes and then suctioned out through the bronchoscope.

Next, 3 study doctors will check how well the mucus in your stent was cleared. If the study doctors think not enough mucus has been cleared from your stent, you will "crossover" into the other study group and receive the other agent to clear your mucus.

Length of Study:

Your participation on the study will be over after you have completed the follow-up visits.

Follow-Up:

At about 7 days, and then again 30 days after your bronchoscopy, you will come to the clinic for a follow-up visit. The following procedures will be performed:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will also be asked about any side effects you may be having.

This is an investigational study. Normal saline and sodium bicarbonate are agents used in bronchoscopies performed in patients with airway stents as standard of care. The comparison of sodium bicarbonate to normal saline to clear mucus from airway stents is considered investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>/= 18 years) with airway stents undergoing bronchoscopy.
2. Patients previously enrolled, but excluded as no stent lumen obstruction from mucus retention identified at earlier enrollment (hence excluded at that enrollment) .

Exclusion Criteria:

1. Patients with history of allergy or adverse reactions to sodium bicarbonate or normal saline.
2. Patients refusing to sign informed written consent for participation in research.
3. Patients with no stent lumen occlusion from mucus impaction as determined at the time of the initial visual bronchoscopic assessment.
4. Previously enrolled patients who completed this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of obstruction resolution as Good or Excellent | Baseline to 7 days
  Response/efficacy of sodium bicarbonate versus normal saline in airway stents graded using scale. Percentage of obstruction resolution (relative to initial stent lumen obstruction by mucus): Good response 51-75% clearance; and Excellent 76 - 100% clearance. The Mantel-Haenszel chi-square test stratified by degree of lumen obstruction at study enrollment used to compare response (good or excellent obstruction resolution) rates between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Jimenez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Website — http://www.mdanderson.org